CLINICAL TRIAL: NCT02072083
Title: Intranasal Dexmedetomidine Versus Intranasal Midazolam-ketamine Combination for Premedication of Pediatric Patients Undergoing Strabismus Surgery
Brief Title: Intranasal Dexmedetomidine vs Midazolam-ketamine Combination for Premedication of Pediatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, müge yüce yıldırım, resident, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2013/381
Record Dates: First submitted 2014-02-15; First posted 2014-02-26 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2014-02

CONDITIONS: Premedication; Oculocardiac Reflex
Keywords: dexmedetomidine; intranasal; strabismus surgery; premedication; oculocardiac reflex
MeSH Terms: interventions — Dexmedetomidine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine (Active Comparator): intranasal 1mcg/kg
  Interventions: Drug: Dexmedetomidine
- ketamine (Active Comparator): intranasal 7,5 mg/kg ketamine and 0,1 mg/kg midazolam
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Dexmedetomidine — via intranasal route 1 mcg/kg
  Other Names: precedex
  Arms: dexmedetomidine
Drug: Ketamine — via intranasal route 7,5 mg/kg ketamine and 0,1 mg/kg midazolam
  Other Names: ketalar
  Arms: ketamine

SUMMARY:
The aim of this study is using intranasal dexmedetomidine versus intranasal midazolam-ketamine combination for premedication and preventing the oculocardiac reflex of pediatric patients undergoing strabismus surgery.

DETAILED DESCRIPTION:
Preanesthetic medication in pediatrics is very helpful in relieving anxiety, fear and psychological trauma due to maternal deprivation. Midazolam and ketamine are commonly used for this purpose. Dexmedetomidine is an alpha 2 -agonist with a more selective action on the alpha 2 adrenoreceptor when administered via the nasal mucosa bioavailability of dexmedetomidine is too high. Intranasal route is an effective way to administer premedication and sedation to children. The oculocardiac reflex is a major complication of pediatric strabismus surgery.

ELIGIBILITY:
Inclusion Criteria:

* the pediatric patients undergoing strabismus surgery
* the pediatric patients between 2-11 years old
* ASA physical status I-II
* the patients whose parents give permission for this study

Exclusion Criteria:

* a known drud allergy or hypersensitive reaction to drugs used
* mental retardation
* cardiac arrhythmia or congenital cardiac disease
* organ disfunction (liver , kidney)
* nasal pathology
* psychotropic treatment

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
the efficacy of premedication on ramsey sedation score | 30 min after premedication
  after drug administration ramsey sedation scale is evaluate every 5 min.

SECONDARY OUTCOMES:
the effects of premedication on oculocardiac reflex | during the surgery
  the heart rate drops the 20% of the resting rate
mask acceptance scale | 30 min after sedation
  The subject's ability to accept the anesthesia mask is measured using the mask acceptance scale.
the parenteral separation anxiety scale | 30 min after sedation
  The response to the child parent separation is assessed and graded according to a 4 point scale at 30 min.

CONTACTS AND LOCATIONS:
Overall Officials: Müge Yüce Yıldırım, resident, Principal Investigator — erciyes univercity
Locations (1):
- Erciyes university hospital, Kayseri, Turkey (Türkiye)